CLINICAL TRIAL: NCT03766126
Title: Phase 1 Study of Lentivirally Transduced T Cells Engineered to Contain Anti-CD123 Linked to TCRζ and 4-1BB Signaling Domains in Subjects With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Lentivirally Redirected CD123 Autologous T Cells in AML
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 831619 (UPCC 35418)
Record Dates: First submitted 2018-12-03; First posted 2018-12-06 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia, Adult; Acute Myeloid Leukemia, Refractory
Keywords: refractory; relapsed; Acute; Myeloid; leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Leukemia | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): CART123 cells; cyclophosphamide; fludarabine
  Interventions: Biological: CART123 cells; cyclophosphamide; fludarabine

INTERVENTIONS:
Biological: CART123 cells; cyclophosphamide; fludarabine — CART123 cells following lymphodepleting chemotherapy in patients with relapsed/refractory AML. Subjects will be treated with a split dosing approach of CART123 cells (10% Day 0; 30% Day 1; 60% Day 2) for Cohort 1a/1b or a single IV administration of CART123 cells for Cohort 2.
  The total dose administered to each subject will be based on body weight obtained at the time of apheresis. Thus, the target total transduced dose, preceded by lymphodepleting chemotherapy, is 1-2x10^6 CART123 cells/kg for Cohort 1a, 5x10^6 CART123 cells/kg for Cohort 1b, or 2x10^6 CART-123 cells/kg for Cohort 2. The protocol-specified minimum acceptable dose for infusion is 1x10^5 CART123 cells/kg.
  Other Names: T Cells Containing Anti-CD123 Signaling Domains

SUMMARY:
Phase 1 open-label study to estimate the safety, manufacturing feasibility, and efficacy of intravenously administered, lentivirally transduced T cells expressing anti-CD123 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ /4-1BB) costimulatory domains in Acute Myeloid Leukemia (AML) subjects.

DETAILED DESCRIPTION:
This is a Phase 1 study to determine the safety, feasibility, and efficacy of CART123 cells following lymphodepleting chemotherapy in patients with relapsed/refractory AML. Subjects will be treated with a split dosing approach of CART123 cells (10% Day 0; 30% Day 1; 60% Day 2) for Cohort 1a/1b or a single IV administration of CART123 cells for Cohort 2.

The total dose administered to each subject will be based on body weight obtained at the time of apheresis. Thus, the target total transduced dose, preceded by lymphodepleting chemotherapy, is 1-2x10^6 CART123 cells/kg for Cohort 1a, 5x10^6 CART123 cells/kg for Cohort 1b, or 2x10^6 CART-123 cells/kg for Cohort 2. The protocol-specified minimum acceptable dose for infusion is 1x10^5 CART123 cells/kg for all cohorts.

It is recommended per routine clinical care, that all subjects with marrow aplasia at Day 28+/-5 undergo allogeneic hematopoietic cell transplantation (alloHCT) as a rescue strategy. If required, this procedure will be performed as part of routine care, outside of the scope of this research study, however subjects will continue to be followed on study. All subjects should therefore have a previously identified stem cell donor in order to participate in this study. Please see Section 6.8 for additional details.

All subjects will be followed monthly for up to 6 months post the first CART123 cell infusion (Day 0). Thereafter subjects will be transitioned into LTFU for up to 15 years post infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age or older
2. Subjects with active acute myeloid leukemia (AML) with no available curative treatment options using currently available therapies. Specifically:

   1. AML that has not achieved a complete remission or morphologic leukemia free state by ELN criteria (Döhner et al., 2017 Blood, 129(4):424-447); partial remission or refractory disease (including primary refractory) are eligible. Or:
   2. AML relapsed following allogeneic stem cell transplantation (including MDS evolved to AML post-allogeneic stem cell transplantation). Note: morphologic relapse is not required; persistent/recurrent disease-associated molecular, phenotypic or cytogenetic abnormalities (measurable residual disease, MRD) at any time after allogeneic HCT is eligible
3. Subjects with relapsed disease after prior transplant must meet one of the following:

   a. Subjects with relapsed disease after prior allogeneic HCT (myeloablative or non-myeloablative) will be eligible if they meet all other inclusion criteria and i. Have no residual donor cells (by STR analysis on 2 occasions separated by at least 1 month), OR: ii. Donor cells are present but there is no active GVHD (>Gr II), subject does not require systemic immunosuppression and is more than 3 months from transplant, and at least 1 month off GVHD prophylaxis.

   b. Subjects with relapsed disease after prior autologous or syngeneic HCT will be eligible if they meet all other inclusion criteria and it has been more than 3 months from transplant.
4. Subjects must have a suitable stem cell donor available who may donate cells in the event the subject needs to undergo an allogeneic HCT. Donor may be matched or mismatched and must be found to be suitable according to the institution's standard criteria; donors must be fully cleared to proceed as the donor.
5. Satisfactory organ functions:

   1. Creatinine ≤ 1.6 mg/dl
   2. ALT/AST must be ≤5 x upper limit of normal unless related to disease
   3. Direct bilirubin or total bilirubin < 2.0mg/dl, unless subject has Gilbert's syndrome (≤3.0 mg/dL);
   4. Left ventricular ejection fraction ≥ 40% as confirmed by ECHO/MUGA
6. ECOG Performance status 0-2.
7. Written informed consent is given.
8. No contraindications for leukapheresis.
9. Subjects of reproductive potential must agree to use acceptable birth control methods (as described in protocol Section 4.3).

Exclusion Criteria:

1. Pregnant or lactating (nursing women) women.
2. Patients with relapsed AML with t(15:17).
3. HIV infection.
4. Active hepatitis B or hepatitis C infection.
5. Concurrent use of systemic steroids or immunosuppressant medications. Recent or current use of inhaled steroids or physiologic replacement with hydrocortisone is not exclusionary. For additional details regarding use of steroids while on study, please see Section 5.5.
6. Any uncontrolled active medical disorder that would preclude participation as outlined.
7. Subjects with signs or symptoms indicative of CNS involvement. A CNS evaluation should be performed as clinically appropriate to rule out CNS involvement.
8. Known history of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
9. Class III/IV cardiovascular disability according to the New York Heart Association Classification (see Appendix 3).
10. Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, and unrelated to leukemia or previous leukemia treatment.
11. Subjects with clinically apparent arrhythmia, or arrhythmias that are not stable on medical management, within 2 weeks of the Screening/Enrollment visit.
12. Patients with any prior history of myeloproliferative neoplasm.
13. Patients with the JAK2 V617F mutation by PCR or next generation sequencing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2033-12-03 (Estimated); Study Completion 2033-12-03 (Estimated)

PRIMARY OUTCOMES:
Safety profile of CART123 cells by monitoring the frequency and severity of adverse events assessed by the National Cancer Institute (NCI) - Common Toxicity Criteria (v5.0) | 5 years
  Assess the safety of CART123 cells in AML subjects following lymphodepletion with cyclophosphamide + fludarabine.
Evaluate the percentage of manufacturing products that do not meet release criteria for vector transduction efficiency, T cell product purity, viability, sterility. | 5 year
  Evaluate the percentage of manufacturing products that do not meet release criteria for vector transduction efficiency, T cell product purity, viability, sterility.

SECONDARY OUTCOMES:
Estimation of CART123 efficacy by evaluation of OS and PFS of subjects at protocol defined intervals which receive at least one infusion of CART123 cells | 15 years
  Estimate the efficacy of at least 1 dose of CART123 cells in AML subjects
Overall Survival (OS) as percent of subjects surviving at protocol defined time points. | 15 years
  Overall survival (OS) and progression-free survival (PFS)
Progression-free survival (PFS) as percent of subjects surviving without disease progression at protocol defined time points | 15 years
Duration of response (DOR) | 15 years
  Duration of response (DOR)
Necessity of rescue bone marrow transplant | 15 years
  Need for rescue allogeneic hematopoietic cell transplantation (alloHCT)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhagwat AS, Torres L, Shestova O, Shestov M, Mellors PW, Fisher HR, Farooki SN, Frost BF, Loken MR, Gaymon AL, Frazee D, Rogal W, Frey N, Hexner EO, Luger SM, Loren AW, Martin ME, McCurdy SR, Perl AE, Stadtmauer EA, Brogdon JL, Fraietta JA, Hwang WT, Siegel DL, Plesa G, Aplenc R, Porter DL, June CH, Gill SI. Cytokine-mediated CAR T therapy resistance in AML. Nat Med. 2024 Dec;30(12):3697-3708. doi: 10.1038/s41591-024-03271-5. Epub 2024 Sep 27. PMID 39333315